CLINICAL TRIAL: NCT01160159
Title: Arterial Microcirculation, Macrocirculation and Thrombophilias
Acronym: MICMAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department of clinical research and development
Other Study IDs: P071012; IDRCB 2008-A01635-50 (Other: AFSSAPS)
Record Dates: First submitted 2010-02-19; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-02

CONDITIONS: Thrombophilia
Keywords: Venous thrombosis; Women; Vasodilatation endothelium-dependent; IMT; Arterial stiffness; Arterial compliance; Capillary density
MeSH Terms: conditions — Thrombophilia; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thrombophilia
  Interventions: Other: Tests
- Healthy volunteers
  Interventions: Other: Healthy volunteers

INTERVENTIONS:
Other: Tests — Arterial parameters
  Groups: Thrombophilia
Other: Healthy volunteers — Arterial parameters and blood test
  Groups: Healthy volunteers

SUMMARY:
Rationale: To analyse the arterial state of women with thrombophilia by techniques studying micro and arterial macrocirculation because of a reported and still discussed increase risk in cardio-vascular events in these women.

Primary objective: To measure endothelium dependent vasodilatation (VDE) in controls and in women with thrombophilia.

DETAILED DESCRIPTION:
There are several papers reporting an increase in the risk of arterial diseases in women with thrombophilia. However these reports remain controversial. In order to gain insight on that issue we propose to study the micro and macrocirculation in women with an history of venous thrombosis or thrombophilia and in controls matched by age.

Design: It is a prospective open transversal trial.

Management of the study: Two groups of 80 women will be compared: healthy volunteers and women with thrombophilia. Following an inclusion consultation where the informed consent will be obtained and inclusion criteria checked, an appointment for the arterial explorations will be given. These explorations will be measurement of endothelium dependent vasodilatation (EDV), capillar density, arterial fitness and compliance and retinogram. There is no follow-up visit.Benefits and risks: the measurement will characterize the arterial state of patients with thrombophilia included in the study.There is no risk in performing these techniques.

Principal criteria: measurement of EDV.

Secondary criteria: capillar density, arterial compliance and stiffness and retinogram.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

  * 18-45 years old women of child bearing age
  * Without any hormonal contraception nor any hormone treatment since at least 3 months
  * Without any arterial risk factors (HTA, diabetes, dyslipemia, obesity, including smoking> 5 cigaret )
  * Patient who have signed an inform consent
  * With no thrombophilia : normal sample for factor V and II mutations
  * Willing to participate to the study
  * Adherent to health insurance
  * Previous Clinical examination
* women with thrombophilia

  * 18-45 years old women of child bearing age
  * Without any hormonal contraception nor any hormone treatment since at least 3 months
  * Without any arterial risk factors (HTA, diabetes, dyslipemia, obesity, including smoking> 5 cigaret )
  * Patient who have signed an inform consent
  * With thrombophilia : normal sample for factor V and II mutations
  * Willing to participate to the study
  * Adherent to health insurance
  * Previous Clinical examination

Exclusion Criteria:

* Women under hormonal contraception or who have stopped it less than 3 months ago
* Women under anticoagulant
* Arterial risk factor : HTA, diabetes, dyslipemia, obesity(BMI>30), including smoking> 5 cigarets ), metabolic syndrome, antiphospholipids/anticoagulant antibody, SLE
* History of coronaropathy or of stroke
* Pregnant women or willing to conceive
* Severe liver disease
* Women of less than 18y or older than 45y
* Severe liver diseases
* Patient not willing to sign up the inform consent
* Patient refusal to participate
* Endometrial cancer
* Unexplored bleeding
* Women not willing to participate or included in another trial
* Woman with another thrombophilic disorder (ATIII, protein C, S, history of VTE without any biological thrombophilic disorder.
* Women with at least one of the following treatment and who cannot stop it 48h before the arterial investigations.
* Gynergen caffeine
* NOCERTONE® oxetorone
* SIBÉLIUM®flunarizine
* VIDORA®indoramine
* SANMIGRAN® 0,50 mg pizotifen
* woman under propranolol AVLOCARDYL® 40 mg *AVLOCARDYL® LP 160 mg

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups of 80 women will be compared: healthy volunteers and women with thrombophilia.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Vasodilatation endothelium-dependent (VDE) | at 2 months max after inclusion

SECONDARY OUTCOMES:
Capillary density | at 2 months max after inclusion
Stiffness and arterial compliance | at 2 months max after inclusion
Analysis of venous and arterial microcirculation using images acquired by retinogram and a specific software | at 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Anne GOMPEL, MD-PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Geneviève PLU-BUREAU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Hotel Dieu - Consultation Gynécologie et d'Hémostase, Paris, France